CLINICAL TRIAL: NCT03554629
Title: A Comparison of Capnography Sampling Lines
Acronym: FRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MDT17063FRS
Record Dates: First submitted 2018-05-01; First posted 2018-06-13 (Actual); Results first posted 2020-12-16 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Capnography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Capnography CO2 Sampling Filterline Performance (Other): Adult volunteer exhaled gas was sampled by 8 different CO2 cannula sampling filterline (CCSF) designs connected to a Capnostream 35 for measurement of CO2 during patient simulated scripted activities in order to assess patient interface design performance to provide a quality gas sample for CO2 partial pressure measurement.
  Interventions: Device: Capnography CO2 cannula sampling Flexiterline (CCSF) designs with supplemental O2

INTERVENTIONS:
Device: Capnography CO2 cannula sampling Flexiterline (CCSF) designs with supplemental O2 — Use of 8 post-market nasal CO2 cannula sampling filterlines; 4 nasal only sampling ports manufactured by Medtronic, Salter, Hudson/Teleflex and FlexiCare) and 4 post-market oral/nasal sampling ports manufactured by Medtronic, Salter, Dispo-Med and Westmed during scripted activity with supplemental O2.

SUMMARY:
This study evaluates the performance of eight (8) cleared capnography carbon dioxide (CO2) sampling filterlines during patient simulated scripted activities when connected to a Medtronic (MDT) dual parameter monitor.

DETAILED DESCRIPTION:
The eight (8) Capnography CO2 Sampling Filterlines (CCSF) have different designs for obtaining a gas sample for CO2 measurement and also for delivering supplemental oxygen (O2).

In this study awake, healthy volunteers will evaluate the 8 CCSF (Capnography CO2 Sampling Filterline) to determine their performance variability in providing a representative exhaled CO2 sample for measurement on the Capnostream 35 dual parameter monitor during scripted activities of closed mouth/open mouth breathing during both high and low respiration rate with supplemental oxygen delivery at 5lpm.

ELIGIBILITY:
Inclusion Criteria:

1. Non-hospitalized adults ≥ 18 years old.
2. Willing and able to give informed consent.

Exclusion Criteria:

1. Lack of an informed consent.
2. Subjects not able to accommodate the proper application of the cannula.
3. Subject not willing or able to comply fully with the study procedures.
4. Subjects with sensitivity to nasal cannula in both nares.
5. Subject with skin allergies to medical adhesives.
6. Subjects with runny nose the day of the study participation.
7. Subject, who in the opinion of the Principal Investigator, should not be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Miner, MD, Principal Investigator — Clinimark, LLC
Locations (1):
- Clinimark LLC, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data will not be shared

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Execution of CIP v 1 enrollment at 6; data not included in results since data inadequate.
  Execution of CIP V2 enrollment was 23 One subject withdrawn before participation due to failure to meet failure to meet criteria of enrollment on the study day (runny nose)
Units Other Than Participants: Nasal/Oral-Nasal Sampling
Groups:
- Eight Capnography CO2 Sampling Filterline Performance: Capnography CO2 Sampling FIlterlines blinded by code name during scripted activities for data analysis.
  All subjects worn all 8 CCSF devices under test for the four study activities.
  1 and 2. Closed mouth breathing with respiration rate of 6 and 24 3 and 4. Open mouth breathing with respiration rate at 6 and 24
Period: Overall Study
Arm/Group | Eight Capnography CO2 Sampling Filterline Performance
Started | 29; 232 Nasal/Oral-Nasal Sampling (8 filterlines per participant for four scripted activities with supplemental oxygen)
Completed | 23; 184 Nasal/Oral-Nasal Sampling (8 filterlines (CCSF) per participate for four scripted activities with supplemental oxygen.)
Not Completed | 6; 48 Nasal/Oral-Nasal Sampling
Not completed — Inadequate data | 6

BASELINE CHARACTERISTICS:
Population: One subject withdrawn before study participation Data on 6 subjects removed due to insufficient data
Groups:
- Capnography CO2 Sampling Filterline: Capnography CO2 Sampling Filterline: Use of up to 8 Capnography CO2 Sampling FIlterlines by blinded code name during scripted activities
Arm/Group | Capnography CO2 Sampling Filterline
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.5 (6.6)

OUTCOME MEASURES:

1. Primary Outcome: Capnography Measured CO2 Waveform Data as a Function of CO2 Cannula Sampling Filterline (CCSF) Stratified by Activity
Description: Comparison of measured end-tidal CO2 (EtCO2), Rebreathing as measured by fractional inspiratory CO2 (FiCO2) as a function the activity for 8 different CCSF designs tested on 23 subjects with supplemental O2 at 5lmp for four activities.
  Device data collected a 20Hz (20 data points/second) for the 3 hours of enrollment.
  Participants lateral lying with head on a pillow with supplemental O2 during each nasal only or open mouth breathing at respiration rate of 6 and 24.
Time Frame: Three hours
Population: Performance of 8 CO2 cannula sampling filterlines (CCSF): 4 filterlines provided nasal only sampling ports and 4 filterlines provided both nasal and oral sampling ports.
  Each of the 8 CCSF was assigned a letter by the investigation site to maintain blinding in data analysis.
  Side-stream capnography measurement via the Capnostream 35
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- EtCO2 During Mouth Closed Breathing Rate of 6: Patient interface to sample gas for EtCO2 capnography measurement under condition of closed mouth and respiration rate of 6 with supplemental O2 at 5lpm.
- FiCO2 During Mouth Closed Breathing Rate of 6: Patient interface to remove stale air when providing a gas sample for capnography measurement of Fractional Inspired CO2 (re-breathing) under condition of closed mouth and respiration rate of 6 with supplemental O2 at 5lpm.
- EtCO2 During Mouth Closed Breathing Rate of 24: Patient interface to sample gas for end tidal CO2 (EtCO2)capnography measurement under condition of closed mouth and respiration rate of 24 with supplemental O2 at 5lpm.
- FiCO2 During Mouth Closed Breathing Rate of 24: Patient interface to remove stale air when providing a gas sample for capnography measurement of Fractional Inspired CO2 (re-breathing) under condition of closed mouth and respiration rate of 24 with supplemental O2 at 5lpm.
- EtCO2 During Mouth Open Breathing Rate of 6: Patient interface to sample gas for end tidal CO2 (EtCO2) capnography measurement under condition of open mouth breathing and respiration rate of 6 with supplemental O2 at 5lpm.
- FiCO2 During Mouth Open Breathing Rate of 6: Patient interface to remove stale air when providing a gas sample for capnography measurement of Fractional Inspired CO2 (re-breathing) under condition of open mouth breathing and respiration rate of 6 with supplemental O2 at 5lpm.
- EtCO2 Mouth Open Breathing Rate of 24: Patient interface to sample gas for capnography measurement under condition of open mouth breathing and respiration rate of 24 with supplemental O2 at 5lpm.
- FiCO2 Mouth Open Breathing Rate of 24: Patient interface to remove stale air when providing a gas sample for capnography measurement of Fractional Inspired CO2 (re-breathing) under condition of open mouth breathing and respiration rate of 24 with supplemental O2 at 5lpm.
Arm/Group | EtCO2 During Mouth Closed Breathing Rate of 6 | FiCO2 During Mouth Closed Breathing Rate of 6 | EtCO2 During Mouth Closed Breathing Rate of 24 | FiCO2 During Mouth Closed Breathing Rate of 24 | EtCO2 During Mouth Open Breathing Rate of 6 | FiCO2 During Mouth Open Breathing Rate of 6 | EtCO2 Mouth Open Breathing Rate of 24 | FiCO2 Mouth Open Breathing Rate of 24
Number analyzed (Participants) | 23 | 23 | 23 | 23 | 23 | 23 | 23 | 23
mmHg
  FlexiCare (Nasal) | 30.6 (7.5) | 0.0 (0.2) | 26.6 (6.2) | 0.2 (0.8) | 20.1 (12.5) | 0.1 (0.2) | 19.1 (10.2) | 0.2 (0.6)
  Hudson RCI /TeleFlex(Nasal) | 13.5 (8.4) | 0.0 (0.0) | 12.3 (6.9) | 0.0 (0.1) | 7.6 (6.6) | 0.0 (0.0) | 7.8 (7.2) | 0.0 (0.0)
  Salter Lab (Nasal) | 30.1 (5.5) | 0.4 (0.8) | 24.1 (5.9) | 1.4 (1.2) | 22.3 (9.2) | 0.2 (0.3) | 19.9 (7.6) | 1.0 (1.1)
  Medtronic Filterline (Nasal) | 32.6 (5.4) | 0.0 (0.0) | 28.1 (5.2) | 0.0 (0.2) | 24.8 (8.3) | 0.0 (0.0) | 22.7 (7.6) | 0.0 (0.0)
  WestMed (Oral/Nasal) | 33.9 (4.8) | 0.5 (0.4) | 29.2 (5.8) | 1.4 (1.5) | 28.0 (8.9) | 0.5 (0.6) | 24.1 (8.1) | 1.2 (1.4)
  Dispo-Med (Oral/Nasal) | 29.9 (7.5) | 0.1 (0.3) | 23.8 (8.2) | 1.4 (0.9) | 23.6 (6.9) | 0.1 (0.2) | 19.3 (7.0) | 1.4 (1.3)
  Salter Lab Oral-Trac (Oral/Nasal) | 29.3 (8.7) | 0.3 (0.5) | 25.0 (6.9) | 0.6 (0.9) | 26.8 (5.2) | 0.2 (0.3) | 23.4 (4.7) | 0.9 (1.1)
  Medtronic Smart Capnoline+(Oral/Nasal) | 32.6 (5.4) | 0.0 (0.0) | 28.8 (4.8) | 0.0 (0.1) | 26.8 (7.4) | 0.0 (0.0) | 24.9 (6.2) | 0.0 (0.1)

2. Secondary Outcome: Average Number of Alarms as a Function of Each Capnography CO2 Cannula Sampling Filterline (CCSF) Stratified by Activity With an Actual Respiration Rate of 24
Description: Gas sample provided by CCSF to the Capnostream 35 for measurement of the partial pressure of CO2 as a function of time.
  The Capnostream 35 Respiration rate algorithm counts the breaths per minute based upon the frequency of a CO2 validated breath waveform.
Time Frame: Three hours
Population: Participant actual Respiration Rate was coached using the Pace Breathing Android App: Version 2.1.
  RR = 6 : Inspiratory Time was 5.0 seconds and Expiratory time was 5.0 seconds No breath alarm is deployed when both RR and EtCO2 are equal to zero. RR = 24: Inspiratory Time was 1.2 seconds and Expiratory time was 1.3 seconds
Measure: Mean (Standard Deviation); unit: Alarms
Groups:
- 20 Second No Breath Alarm With Actual Respiration Rate of 24: When actual respiration rate was 24 breaths per minute
  CO2 derived RR from the gas sample provide by the CO2 Cannula Sampling Filterline (CCSF)
- 30 Second No Breath Alarm With Actual Respiration Rate of 24: When actual respiration rate was 24.
  CO2 derived RR from the gas sample provide by the CO2 Cannula Sampling Filterline (CCSF)
- 15 Second LOW RR 18 Alarm With Actual Respiration Rate of 24; 15 Second LOW RR 6 Alarm With Actual Respiration Rate of 24; 30 Second LOW RR 6 With Actual Respiration Rate of 24: False Low RR for 15 - 29 seconds with patient interface gas sample for capnography derived respiration measurement under condition of subject respiration rate of 24 with supplemental O2 at 5lpm.
- 30 Second LOW RR 18 With Actual Respiration Rate of 24: False Low RR for 15- 29 seconds with CCSF gas sample for capnography measurement.
Arm/Group | 20 Second No Breath Alarm With Actual Respiration Rate of 24 | 30 Second No Breath Alarm With Actual Respiration Rate of 24 | 15 Second LOW RR 18 Alarm With Actual Respiration Rate of 24 | 30 Second LOW RR 18 With Actual Respiration Rate of 24 | 15 Second LOW RR 6 Alarm With Actual Respiration Rate of 24 | 30 Second LOW RR 6 With Actual Respiration Rate of 24
Number analyzed (Participants) | 23 | 23 | 23 | 23 | 23 | 23
Alarms
  FlexiCare (Nasal) | 0.17 (0.53) | 0.13 (0.40) | 0.35 (0.57) | 0.30 (0.51) | 0.17 (0.38) | 0.15 (0.36)
  Hudson/TeleFlex (Nasal) | 0.20 (0.40) | 0.13 (0.34) | 0.74 (0.53) | 0.63 (0.57) | 0.52 (0.51) | 0.50 (0.51)
  Salter Labs (Nasal) | 0.02 (0.15) | 0.02 (0.15) | 0.37 (0.61) | 0.22 (0.47) | 0.13 (0.34) | 0.04 (0.21)
  Medtronic CO2 (Nasal) | 0.02 (0.15) | 0.02 (0.15) | 0.17 (0.38) | 0.11 (0.31) | 0.13 (0.40) | 0.07 (0.25)
  WestMed (Oral/Nasal) | 0.04 (0.29) | 0.04 (0.29) | 0.13 (0.34) | 0.11 (0.31) | 0.09 (0.28) | 0.09 (0.28)
  DispoMed (Oral/Nasal) | 0.04 (0.21) | 0.04 (0.21) | 0.37 (0.53) | 0.28 (0.46) | 0.20 (0.45) | 0.15 (0.36)
  Salter Oral-Trac (Oral/Nasal) | 0.02 (0.15) | 0.02 (0.15) | 0.22 (0.47) | 0.11 (0.31) | 0.13 (0.40) | 0.07 (0.25)
  Medtronic Smart CapnoLine Plus (Oral/Nasal) | 0.00 (0.00) | 0.00 (0.00) | 0.09 (0.28) | 0.09 (0.28) | 0.04 (0.21) | 0.04 (0.21)

3. Secondary Outcome: Average Number of Alarms as a Function of Each Capnography CO2 Cannula Sampling Filterline (CCSF) Stratified by Activity With an Actual Respiration Rate of 6
Description: as for outcome 2
Time Frame: Three hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Alarms
Groups:
- 20 Second No Breath Alarm With Actual Respiration Rate of 6: When actual respiration rate was 6 breaths per minute
  CO2 derived RR from the gas sample provide by the CO2 Cannula Sampling Filterline (CCSF)
- 30 Second No Breath Alarm With Actual Respiration Rate of 6: When actual respiration rate was 6 .
  CO2 derived RR from the gas sample provide by the CO2 Cannula Sampling Filterline (CCSF)
- 15 Second LOW RR 4 Alarm With Actual Respiration Rate of 6: False Low RR for 15 - 29 seconds with patient interface gas sample for capnography derived respiration measurement under condition of subject respiration rate of 24 with supplemental O2 at 5lpm.
- 30 Second LOW RR 4 With Actual Respiration Rate of 6: False Low RR for 15- 29 seconds with CCSF gas sample for capnography measurement.
Arm/Group | 20 Second No Breath Alarm With Actual Respiration Rate of 6 | 30 Second No Breath Alarm With Actual Respiration Rate of 6 | 15 Second LOW RR 4 Alarm With Actual Respiration Rate of 6 | 30 Second LOW RR 4 With Actual Respiration Rate of 6
Number analyzed (Participants) | 23 | 23 | 23 | 23
Alarms
  FlexiCare (Nasal) | 0.13 (0.34) | 0.09 (0.28) | 0.24 (0.43) | 0.22 (0.42)
  Hudson/TeleFlex (Nasal) | 0.30 (0.55) | 0.24 (0.48) | 0.54 (0.55) | 0.43 (0.50)
  Salter Labs (Nasal) | 0.11 (0.31) | 0.07 (0.25) | 0.11 (0.31) | 0.09 (0.28)
  Medtronic CO2 (Nasal) | 0.07 (0.25) | 0.07 (0.25) | 0.13 (0.34) | 0.09 (0.28)
  WestMed (Oral/Nasal) | 0.02 (0.15) | 0.02 (0.15) | 0.07 (0.33) | 0.04 (0.21)
  DispoMed (Oral/Nasal) | 0.04 (0.21) | 0.02 (0.15) | 0.11 (0.31) | 0.07 (0.25)
  Salter Oral-Trac (Oral/Nasal) | 0.04 (0.21) | 0.04 (0.21) | 0.11 (0.31) | 0.07 (0.25)
  Medtronic Smart CapnoLine Plus (Oral/Nasal) | 0.0 (0.0) | 0.0 (0.0) | 0.07 (0.25) | 0.07 (0.25)

ADVERSE EVENTS:
Time Frame: 3 hours
Description: Hypoxemia
Groups:
- FlexiCare (Nasal); Hudson RCI /TeleFlex(Nasal); Salter Lab (Nasal); Medtronic Filterline (Nasal); WestMed (Oral/Nasal) RCI /TeleFlex(Nasal); Dispo-Med (Oral/Nasal); Salter Lab Oral-Trac (Oral/Nasal); Medtronic Smart Capnoline+(Oral/Nasal): 8 Capnography CO2 Sampling FIlterlines blinded by code name during scripted activities with supplemental oxygen at 5lpm for each participant.
  Adverse event Conditions that required a stop of the procedures until SpO2 > 90% were the following
Arm/Group | FlexiCare (Nasal) | Hudson RCI /TeleFlex(Nasal) | Salter Lab (Nasal) | Medtronic Filterline (Nasal) | WestMed (Oral/Nasal) RCI /TeleFlex(Nasal) | Dispo-Med (Oral/Nasal) | Salter Lab Oral-Trac (Oral/Nasal) | Medtronic Smart Capnoline+(Oral/Nasal)
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29 | 0/29 | 0/29 | 0/29 | 0/29 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/29 | 0/29 | 0/29 | 0/29 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 2/29 | 1/29 | 0/29 | 1/29 | 2/29 | 0/29 | 0/29 | 1/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FlexiCare (Nasal) (N=29) | Hudson RCI /TeleFlex(Nasal) (N=29) | Salter Lab (Nasal) (N=29) | Medtronic Filterline (Nasal) (N=29) | WestMed (Oral/Nasal) RCI /TeleFlex(Nasal) (N=29) | Dispo-Med (Oral/Nasal) (N=29) | Salter Lab Oral-Trac (Oral/Nasal) (N=29) | Medtronic Smart Capnoline+(Oral/Nasal) (N=29)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 — Low Oxygenation with SpO2 < 90% via finger pulse Oximeter Supplemental O2 at 5lpm Occurred with Open Mouth Breathing at RR = 6
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 | 0 | 1 (1) | 0 | 0 | 1 (1) — Low Oxygenation with SpO2 < 90% via finger pulse Oximeter Supplemental O2 at 5lpm Occurred with Open Mouth Breathing at RR = 24
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 — Low Oxygenation with SpO2 < 90% via finger pulse Oximeter Supplemental O2 at 5lpm Occurred with Closed Mouth Breathing at RR = 6

LIMITATIONS AND CAVEATS:
Strategy to test four simulated patient activities that would most likely effect a quality gas sample for measurement of CO2 partial pressure was selected to maintain active enrollment to three hours .

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/29/NCT03554629/SAP_001.pdf
  • Study Protocol (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT03554629/Prot_002.pdf